CLINICAL TRIAL: NCT06352814
Title: Impact of an Activities-based Locomotor Training Program Versus Traditional Physical Therapy in Children With Cerebral Palsy on Activity, Participation, and Neurophysiological Adaptations
Brief Title: Activities-based Locomotor Training Program Versus Traditional Physical Therapy in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Megan Flores, Clinical Associate Professor, Baylor University
Other Study IDs: 1977152
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; children; activities-based locomotor training; neuroplasticity
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ABLT vs traditional PT: Activities-based locomotor training is implemented through a combination of partial body weight supported treadmill training, overground walking, and play-based activities.
  Interventions: Other: Activities-based locomotor training (physical therapy)

INTERVENTIONS:
Other: Activities-based locomotor training (physical therapy) — AB-LT is implemented through a combination of partial body weight supported treadmill training, overground walking, and play-based activities.

SUMMARY:
The purpose of this study is to investigate the impact of an intensive activities-based locomotor training program as compared to traditional physical therapy on activity, participation, and central and peripheral neurophysiological adaptation in children with cerebral palsy.

DETAILED DESCRIPTION:
Observational research will be performed to assess the change in outcome measure scores over time among participants after the AB-LT intervention. Outcome measures will be obtained 4 times, occurring every 3 weeks over a period of 9 weeks: pre-intervention, post-intervention, pre-traditional therapy, and post-traditional therapy. A washout period of 3 weeks will occur between the AB-LT intervention and traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP
* Between the ages of 2 to 12 years.
* Enrolled in a 3-week AB-LT program and/or participate in traditional physical therapy.

Exclusion Criteria:

* Surgery or botulinum toxin injections in the previous 6 months
* Uncontrolled epilepsy or cardiovascular disease.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Community sample (central Texas)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 (GMFM) | 9 weeks
  Gross Motor Function Measure-66: Items scored on 0-3 scale. Minimum value: 0. Maximum value: 99. Higher scores indicate better outcome.
Pediatric Neuromuscular Recovery Scale (PedsNRS) | 9 weeks
  Pediatric Neuromuscular Recovery Scale: Each of the 13 items on the Peds NRS have 12 phases. Each item is scored on a 12-point scale, with one point allocated to each phase of the item. The age-appropriate item cards instruct the rater to begin at a designated "start phase" indicated by a bold box around the phase within the 12 phases on each card. If the child cannot perform the movement as listed in the start phase (which may be midway through the card), the rater starts at the beginning of the item card and assesses the child's performance at the first phase for that item. The rater continues sequentially through the 12 phases on the card until the child is unable to perform a phase. The rater scores the highest phase achieved by the child and moves on to the next item card, through all 13 items. Items are then summed into a summary Peds NRS score using an algorithm.
Pediatric Evaluation of Disability Inventory (PEDI-CAT) | 9 weeks
  Parent questionnaire about child's mobility and activitiies of daily living. Normative Standard Scores: provided as age percentiles and T-scores Scaled Scores (criterion scores): 20-80 scale.
Pediatric Quality of Life Inventory CP Module (PedsQL-CP) | 9 weeks
  For each of the 4 domains, in addition to scaled scores, normative standard scores (provided as T-scores and age percentiles) are calculated. Normative scores describe the child's performance in comparison to other children of the same age (in one year intervals). For T-scores, the mean for each age group is 50, with a standard deviation of 10 (same format used for normative scores in the original PEDI). Typically, T-scores between 30 and 70 (i.e. mean ± 2 standard deviations) are considered within the expected range for age. Scores below 30 indicate decreased functional ability compared to what is typically expected for that age range. Scores above 70 indicate scores above what is typically expected for that age range. Higher scores indicate better outcome.
Functional near-infrared spectroscopy | 9 weeks
  Non-invasive, continuous wave functional near-infrared spectroscopy using an OctaMon+ (Artinis Medical Systems, Lieden, Netherlands) to track oxygenation status.
Electromyography | 9 weeks
  Electrodes will measure electrical activity in response to reflex stimulation of the muscle of the dominant limbs.
ActiGraph sensors | 9 weeks
  Activity performance will be measured using ActiGraph accelerometers, which are motion sensors worn as a bracelet around the rist designed to detect movement when worn. They have excellent inter-instrument reliability (ICC = 0.98). Physical activity data will be expressed in average counts per minute (CPM) on the basis of the vector magnitude of the triaxial accelerometer. In general, higher average CPM represents a more active child.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Flores, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No